CLINICAL TRIAL: NCT03872388
Title: Atorvastatin in Triple-Negative Breast Cancer (TNBC) Patients Who Did Not Achieve a Pathologic Complete Response (pCR) After Receiving Neoadjuvant Chemotherapy, a Multicenter Pilot Study
Brief Title: Atorvastatin in Treating Patients With Stage IIb-III Triple Negative Breast Cancer Who Did Not Achieve a Pathologic Complete Response After Receiving Neoadjuvant Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0550; NCI-2019-00004 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0550 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Estrogen Receptor Negative; HER2/Neu Negative; Inflammatory Breast Carcinoma; Progesterone Receptor Negative; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Atorvastatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (atorvastatin) (Experimental): Patients receive standard of care atorvastatin PO QD for up to 24 months.
  Interventions: Drug: Atorvastatin
- Group II (capecitabine) (Active Comparator): Patients not eligible to receive atorvastatin, will be enrolled into non-statin observation group with/without capecitabine treatment.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Atorvastatin — Patients will receive Atorvastatin per ASCVD guidelines dosed as either a moderate intensity (20mg/day) or high intensity statin (80mg/day). Tablets are available in either 20mg or 80mg and will be dispensed as per standard of care for up to 24 months as part of the study.
  Patients may also receive capecitabine concurrently with Atorvastatin per physician discretion as standard of care. Standard of care dosing of Capecitabine is a 21 day cycle consisting 14 days on and 7 days off. The starting dosing will be per physician discretion, but may be up to 2500mg/m2 per day.
  Arms: Group I (atorvastatin)
Drug: Capecitabine — Patients not eligible to receive atorvastatin in group II will be enrolled into non-statin observation group with/without capecitabine treatment. Capecitabine administration will be dosed as per standard of care. Standard of care dosing of Capecitabine is a 21 day cycle consisting 14 days on and 7 days off. The starting dosing will be per physician discretion, but may be up to 2500mg/m2 per day.
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Group II (capecitabine)

SUMMARY:
This phase II trial studies how well atorvastatin works in treating patients with stages IIb-III triple negative breast cancer who did not achieve a pathologic complete response to neoadjuvant chemotherapy. Pathologic complete response is the lack of all signs of cancer in tissue samples removed during surgery after upfront chemotherapy. Atorvastatin is used for the treatment of high cholesterol and may reduce the risk of triple negative breast cancer from coming back. Triple-negative breast cancer is a type of breast malignancy that is comprised of cancer cells that do not have estrogen receptors, progesterone receptors, or large amounts of HER2/neu protein. Patients with TNBC do not have established systemic therapies such as anti-estrogens or HER2-targeting agents to reduce recurrence after surgery, and residual cancer found at surgery is associated with higher relapse rate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients with undetectable circulating tumor cells (CTCs) at 6 months in patients with stage IIB/III triple negative breast cancer (TNBC) who did not achieve a pathologic complete response a (pCR) or Residual Cancer Burden-I (RCB-I) after receiving neoadjuvant chemotherapy (NAC) with and without atorvastatin therapy.

SECONDARY OBJECTIVES:

I. To determine if baseline fasting lipid profile level (low density lipoprotein cholesterol [LDL-C]) and/or change in serum lipid levels are a predictive biomarker of change in the proportion of patients with CTCs.

II. To assess effect of biomarkers on atorvastatin treatment response, defined as CTCs, circulating tumor deoxyribonucleic acid (DNA) (ctDNA), erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), serum Interleukin-6 (IL-6) and other inflammatory cytokines, for the purpose of identifying the optimal patient population for future larger scale adjuvant studies.

III. To determine if baseline fasting lipid profile level (LDL-C) and/or change in serum lipid levels are associated with 2-year relapse free survival (RFS) rate.

IV. To determine if baseline CRP and/or change in serum lipid levels are a predictive biomarker of change in the proportion of patients with CTCs.

V. To determine if baseline C-reactive protein (CRP) and/or change in CRP are associated with 2-year RFS rate.

VI. To determine if baseline absolute number of CTCs and/or CTC change are associated with 2-year RFS rate.

VII. To estimate the 2-year RFS rate of patients with TNBC who did not achieve pCR with and without atorvastatin therapy.

VIII. To describe the toxicity and adverse events profile of atorvastatin treatment when given concurrently with standard doses of radiotherapy to the chest wall and regional nodes.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation between multiplexed imaging biomarkers in the normal or tumor tissue taken at the time of surgery, and response to atorvastatin-induced CTC changes or with measured outcomes.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients receive standard of care atorvastatin orally (PO) once daily (QD) for up to 24 months. A physical exam is performed, and blood drawn at 3, 6, 12, 18 and 24 months after starting standard of care treatment or at any time the disease appears to get worse.

GROUP II: Patients not eligible to receive atorvastatin, will be enrolled into non-statin observation group with/without capecitabine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial
* Diagnosis of TNBC (including patients with a clinical diagnosis of triple negative inflammatory breast cancer)
* Has histological confirmation of breast carcinoma
* Have stage IIB or III disease as defined by the American Joint Committee on Cancer version 7 or 8
* Has confirmed TNBC, defined as having estrogen and progesterone receptor < 10% positivity by immunohistochemistry (IHC) and HER2 normal, which is 0 or 1+ by IHC and negative by fluorescence in situ hybridization (FISH) if performed or HER2 2+ by IHC and negative by FISH or HER2 negative by FISH if IHC is not performed
* Received neoadjuvant chemotherapy and did not achieve pCR nor had an RCB-I (we will enroll patients with an RCB-II or RCB-III) following neoadjuvant chemotherapy. Since the RCB index has not been validated in IBC, any amount of residual disease will be allowed. pCR is defined as: a) the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current American Joint Committee on Cancer [AJCC] staging system). Or b) the absence of residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0 ypN0 in the current AJCC staging system)
* Has a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >=100,000 /mcL
* Hemoglobin (Hgb) >= 8 g/dL
* Creatinine levels < 2.0 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN
* Subjects of childbearing potential should be willing to use effective methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of study drug; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; effective methods of birth control include 1). Use of hormonal birth control methods: pills, shots/injections, implants (placed under the skin by a health care provider), or patches (placed on the skin); 2). Intrauterine devices (IUDs); 3). Using 2 barrier methods (each partner must use 1 barrier method) with a spermicide. Males must use the male condom (latex or other synthetic material) with spermicide. Females must choose either a diaphragm with spermicide, or cervical cap with spermicide, or a sponge (spermicide is already in the contraceptive sponge)
* Within 3 months from completion of definitive surgery after neoadjuvant chemotherapy
* Willing to take statin for minimum of two years

Exclusion Criteria:

* Has not recovered from adverse events due to prior therapies, i.e. monoclonal antibody, chemotherapy, targeted small molecule therapy, radiation therapy, or surgery

  * Note: Subjects with =< grade 2 neuropathy, alopecia and general disorders and administration site conditions are an exception to this criterion and may qualify for the study
* Has a known malignancy (other than breast cancer) except basal cell carcinoma or squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known psychiatric or substance abuse disorders and assessed by attending physician that would interfere with cooperation with the requirements of the trial
* Has received prior therapy with a statin within past 6 months or is currently receiving statin therapy; patients who previously received a statin more than 6 months prior to beginning study therapy and who discontinued treatment for reasons other than severe toxicity or allergic reaction are eligible
* Is currently receiving another anti-lipidemic agent other than statin: fibric acid derivatives (i.e. fenofibrate, gemfibrozil), bile acid sequestrants (i.e. cholestyramine, colestipol), ezetimibe, niacin, lovaza (omega-3-acid ethyl esters), red yeast rice, orlistat, phytosterol, and lomitapide
* Known hypersensitivity to statin or any component of the formulation
* Active liver disease or unexplained persistent elevations of serum transaminases, defined as elevated transaminases > 3 x ULN on at least 2 separate occasions 1 week apart
* Pregnancy or women who may become pregnant and not on acceptable form of contraception; lactating women
* Has evidence of distant metastasis
* Record of myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Chronic steroid use as this may prevent any immunomodulatory roles of statin treatment, defined as anticipating need of supraphysiologic dose of steroids for at least 12 weeks while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Barcenas, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Banner - MD Anderson Cancer Center, Gilbert, Arizona
  - Banner - MD Anderson Cancer Center -Northern Colorado, Greeley, Colorado
  - Piedmont Healthcare, Atlanta, Georgia
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2019- May 2022. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 6 participants were accrued and assessed for eligibility and 4 patients were assigned to the cohort.
Groups:
- Cohort 1a: Atorvastatin treatment starting at the beginning of radiation. No xeloda.
- Cohort 1b: No Atorvastatin treatment, assessment before starting radiation, no xeloda.
- Cohort 2a: Atorvastatin treatment after xeloda but starting concurrently with radiation.
- Cohort 2b: No atorvastatin treatment, assessment after xeloda but prior to radiation.
- Cohort 3a: Atorvastatin treatment after radiation and xeloda are complete, with optional pre-xeloda blood draw.
- Cohort 3b: No atorvastatin treatment, assessment after radiation and xeloda are complete, with optional pre-xeloda timepoint
- Cohort 4a: Atorvastatin treatment, after xeloda +/- radiation, enrolled after all other therapies are complete.
- Cohort 4b: No atorvastatin treatment, assessment after xeloda +/- radiation, enrolled after all other therapies are complete.
Period: Overall Study
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 6 participants were accrued and assessed for eligibility and 4 patients were assigned to the cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  |  |  |  |  | 0 | 0 | 0
  Between 18 and 65 years |  |  |  |  |  |  | 2 | 2 | 4
  >=65 years |  |  |  |  |  |  | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  |  |  |  | 2 | 2 | 4
  Male |  |  |  |  |  |  | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  |  |  |  |  | 0 | 0 | 0
  Not Hispanic or Latino |  |  |  |  |  |  | 2 | 2 | 4
  Unknown or Not Reported |  |  |  |  |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  |  |  |  | 0 | 0 | 0
  Asian |  |  |  |  |  |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  | 0 | 0 | 0
  Black or African American |  |  |  |  |  |  | 0 | 0 | 0
  White |  |  |  |  |  |  | 2 | 2 | 4
  More than one race |  |  |  |  |  |  | 0 | 0 | 0
  Unknown or Not Reported |  |  |  |  |  |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  |  |  |  |  | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportions of Patients With Undetectable Circulating Tumor Cells (CTC)
Description: Estimate the proportion of patients with undetectable circulating tumor cells (CTCs) at 6 months in patients with stage IIB/III TNBC who did not achieve a pCR or Residual Cancer Burden-I (RCB-I) after receiving neoadjuvant chemotherapy (NAC) with and without atorvastatin therapy.
Time Frame: At 6 months
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Fasting Lipid Profile Level (Low Density Lipoprotein Cholesterol [LDL-C]) and/or Change in Serum Lipid Levels
Description: Determine if baseline fasting lipid profile level (LDL-C) and/or change in serum lipid levels are a predictive biomarker of change in the proportion of patients with CTCs.
Time Frame: Baseline up to 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Biomarkers on Atorvastatin Treatment Response
Description: Assess effect of biomarkers on atorvastatin treatment response, defined as CTCs, circulating tumor DNA (ctDNA), erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), serum Interleukin-6 (IL-6) and other inflammatory cytokines, for the purpose of identifying the optimal patient population for future larger scale adjuvant studies.
Time Frame: Up to 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Fasting Lipid Profile Level (LDL-C) and 2-year RFS Rate
Description: Fasting lipid profile level (LDL-C) and 2-year RFS rate
Time Frame: Baseline up to 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Baseline C-reactive Protein (CRP) and/or Change in Serum Lipid Levels
Description: Determine if baseline CRP and/or change in serum lipid levels are a predictive biomarker of change in the proportion of patients with CTCs.
Time Frame: Baseline up to 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: CTCs and 2-year RFS Rate
Description: Determine if baseline absolute number of CTCs and/or CTC change are associated with 2-year RFS rate.
Time Frame: Baseline up to 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Recurrence-free Survival (RFS)
Description: Estimate the 2-year RFS rate of patients with TNBC who did not achieve pCR with and without atorvastatin therapy.
Time Frame: At 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events, grade and relationship will be tabulated by treatment arms.
Time Frame: Up to 24 months
Population: Only 1 patient who was treated with atorvastatin came for any follow up appointments, however she missed the 6 month timepoint which is the primary end-point of the study. Therefore she was deemed inevaluable. One other treated patient started treatment and died before the 3 month follow up visit, and hence no data was obtained on any patients for cohort 1-3.
Measure: Number; unit: events
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
events
  Grade 1 |  |  |  |  |  |  | 4 | 12
  Grade 2 |  |  |  |  |  |  | 0 | 3

9. Secondary Outcome: C-reactive Protein (CRP) and 2-year RFS Rate
Description: Determine if baseline C-reactive protein (CRP) and/or change in CRP are associated with 2-year RFS rate.
Time Frame: Baseline up to 2 years
Population: Data were not collected.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were captured from the time the patient signs consent until 24 months follow-up was completed or the patient's disease progressed.
Description: All SAEs, expected or unexpected regardless of attribution. The NCI-CTC version 4.0 will be used to grade all AEs.
Arm/Group | Cohort 1a | Cohort 1b | Cohort 2a | Cohort 2b | Cohort 3a | Cohort 3b | Cohort 4a | Cohort 4b
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=0) | Cohort 1b (N=0) | Cohort 2a (N=0) | Cohort 2b (N=0) | Cohort 3a (N=0) | Cohort 3b (N=0) | Cohort 4a (N=2) | Cohort 4b (N=2)
Back Pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | NA | 1 | 1
Breast pain (Reproductive system and breast disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Heart rate increased (Cardiac disorders) | NA | 0 | NA | NA | NA | NA | 0 | 1
Conjunctivitis infective (Infections and infestations) | NA | NA | NA | NA | NA | NA | 0 | 1
Dizziness (Nervous system disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | NA | NA | NA | 1 | 0
Gait disturbance (General disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Headache (Nervous system disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Hypertension (Vascular disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Lymphedema (Vascular disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Pain (General disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Palpitations (Cardiac disorders) | NA | NA | NA | NA | NA | NA | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | NA | NA | NA | NA | NA | 1 | 0
Skin infection (Infections and infestations) | NA | NA | NA | NA | NA | NA | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | NA | NA | NA | 0 | 1
Upper respiratory infection (Infections and infestations) | NA | NA | NA | NA | NA | NA | 0 | 1
Urinary tract infection (Infections and infestations) | NA | NA | NA | NA | NA | NA | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT03872388/Prot_SAP_000.pdf